CLINICAL TRIAL: NCT02873754
Title: Mobile Health Intervention to Help Low-Income Smokers Quit Smoking and Increase Physical Activity
Brief Title: Smoking Treatment and Exercise Program for Underserved Populations (STEP UP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00074576
Record Dates: First submitted 2016-08-17; First posted 2016-08-19 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-06

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Bupropion; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STEP UP (Experimental): STEP UP is an intervention that combines evidence-based telephone cognitive behavioral counseling for smoking cessation, access to nicotine replacement therapy (NRT; including transdermal nicotine patch and either nicotine polacrilex or nicotine lozenge) and bupropion, and intensive mobile contingency management behavioral therapy administered via a smart-phone based application.
  Interventions: Behavioral: Cognitive Behavioral Counseling; Behavioral: Mobile Contingency Management; Drug: Bupropion; Drug: Transdermal nicotine patch; Drug: Nicotine polacrilex; Drug: Nicotine lozenge

INTERVENTIONS:
Behavioral: Cognitive Behavioral Counseling — Participants will receive five cognitive-behavioral counseling sessions designed to improve rates of smoking cessation, enhance relapse prevention, and increase physical activity.
Behavioral: Mobile Contingency Management — Participants will be asked to provide video recordings of themselves taking carbon monoxide readings in order to confirm smoking abstinence. They will also be asked to wear a fitness tracker to monitor physical activity (i.e., steps walked). Participants are provided monetary reward for videos that suggest smoking abstinence, and for fitness tracker readings that suggest increased physical activity.
Drug: Bupropion — All participants who are medically eligible will be prescribed bupropion, which they will start two weeks prior to their quit day. Dosage will be 150 mg/daily for days 1-7 and 300 mg/daily (administered in two daily doses) until the 6-month follow-up.
  Other Names: Zyban
Drug: Transdermal nicotine patch — Initiated at smoking quit date; 7 mg to 21 mg patch depending on amount smoked by participant
Drug: Nicotine polacrilex — Nicotine gum will be initiated at smoking quit date; 4 mg dose administered as needed
  Other Names: Nicotine gum; nicorette
Drug: Nicotine lozenge — Nicotine lozenge will be initiated at smoking quit date; 4 mg dose administered as needed

SUMMARY:
This project proposes to evaluate the feasibility, acceptability, and efficacy of a mobile intervention to target smoking-cessation and increase physical activity among low-income persons. The intervention is called Smoking Treatment and Exercise Program for Underserved Populations (STEP UP).

DETAILED DESCRIPTION:
This pilot project proposes to evaluate the feasibility, acceptability, and efficacy of a mobile intervention to target smoking-cessation and physical activity among low-income persons. The intervention, named Smoking Treatment and Exercise Program for Underserved Populations (STEP UP), combines a smartphone-based contingency-management application (app), which provides monetary reinforcement for smoking abstinence and physical activity, 5 weeks of telephone-based cognitive-behavioral therapy (CBT) to prevent relapse, nicotine replacement pharmacotherapy, and text-messaging to support physical-activity goals. Participants are given a smartphone, a compact carbon-monoxide (CO) monitor, with which recency of smoking can by determined, and a Garmin Vivosmart wristband step-tracker. Twice a day at semi-random intervals, participants are prompted by the app to submit a video of themselves blowing into the CO monitor. Monetary reinforcement is then immediately provided contingent upon a below-threshold CO reading. The app also continuously syncs with the Garmin step-tracker, providing supportive messaging and bonus incentives-namely doubled reinforcement for smoking abstinence among participants who meet personalized daily step goals. The expected outcome of the project is to provide information to evaluate the efficacy of an innovative approach in preparation for a subsequent larger clinical trial that builds upon the capabilities of mHealth technology to reduce the prevalence of smoking among low income smokers.

ELIGIBILITY:
Inclusion Criteria:

* current household income less than twice the federal poverty guidelines (Finer & Henshaw, 2006; for instance, someone from a family of 4 must have a household income less than $48,500 to be eligible)
* currently smoke >10 cigarettes a day
* smoking for at least the past year
* can speak and write fluent conversational English
* are 18-70 years of age
* are willing to make an attempt to quit smoking and increase physical activity

Exclusion Criteria:

* inability to walk
* expected to have unstable medication regimen during the study
* currently receiving non-study behavioral treatment for smoking
* myocardial infarction in the past 6 months
* contraindication to nicotine replacement therapy (NRT) or bupropion with no medical clearance
* exclusive use of other forms of nicotine such as cigars, pipes, e-cigarettes, or chewing tobacco
* current pregnancy
* current imprisonment or psychiatric hospitalization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dennis, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- STEP UP: STEP UP is an intervention that combines evidence-based telephone cognitive behavioral counseling for smoking cessation, access to nicotine replacement therapy (NRT; transdermal nicotine patch and either nicotine polacrilex or nicotine lozenge) and bupropion, and intensive mobile contingency management behavioral therapy administered via smart-phone.
  Cognitive Behavioral Counseling: Participants will receive five cognitive-behavioral counseling sessions designed to improve rates of smoking cessation, enhance relapse prevention, and increase physical activity.
  Mobile Contingency Management: Participants will be asked to provide video recordings of themselves taking carbon monoxide readings in order to confirm smoking abstinence. They will also be asked to wear a fitness tracker to monitor physical activity (i.e., steps walked). Participants are provided monetary reward for videos that suggest smoking abstinence, and for fitness tracker readings that suggested activity.
Period: Overall Study
Arm/Group | STEP UP
Started | 11
Completed | 5
Not Completed | 6
Not completed — Lost to Follow-up | 5
Not completed — Couldn't complete study procedures | 1

BASELINE CHARACTERISTICS:
Groups:
- STEP UP: STEP UP is an intervention that combines evidence-based telephone cognitive behavioral counseling for smoking cessation, access to nicotine replacement therapy (NRT; transdermal nicotine patch and either nicotine polacrilex or nicotine lozenge) and bupropion, and intensive mobile contingency management behavioral therapy administered via smart-phone.
  Cognitive Behavioral Counseling: Participants will receive five cognitive-behavioral counseling sessions designed to improve rates of smoking cessation, enhance relapse prevention, and increase physical activity.
  Mobile Contingency Management: Participants will be asked to provide video recordings of themselves taking carbon monoxide readings in order to confirm smoking abstinence. They will also be asked to wear a fitness tracker to monitor physical activity (i.e., steps walked). Participants are provided monetary reward for videos that suggest smoking abstinence, and for fitness tracker readings that suggest activity.
Arm/Group | STEP UP
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.45 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Self-report Prolonged Abstinence From Smoking
Description: Participants will be asked to report on smoking since two weeks past quit date. Prolonged abstinence is defined as continued abstinence from smoking beginning at 2 weeks post-quit.
Time Frame: 6 month follow up
Population: 5 participants were withdrawn from analyses because they were lost to contact before study completion. One was withdrawn by the PI because he couldn't perform study procedures.
Measure: Count of Participants; unit: Participants
Groups:
- STEP UP: STEP UP combines the following:
  Cognitive Behavioral Counseling: Participants received 5 cognitive-behavioral counseling sessions designed to improve rates of smoking cessation, enhance relapse prevention, and increase physical activity.
  Mobile Contingency Management via smart-phone: Participants provided video recordings of themselves taking carbon monoxide readings to confirm smoking abstinence. They will also wore a fitness tracker to monitor steps walked. Participants were provided monetary reward for smoking abstinence and increased physical activity.
  Bupropion: Dosage will be 150 mg/daily for days 1-7 and 300 mg/daily (administered in two daily doses).
  Transdermal nicotine patch: Initiated at smoking quit date; 7 mg to 21 mg patch.
  Nicotine polacrilex or lozenge: Nicotine gum or lozenge; 4 mg dose administered as needed.
Arm/Group | STEP UP
Number analyzed (Participants) | 5
Participants | 3

2. Primary Outcome: Number of Participants Whose Prolonged Abstinence is Bio-verified
Description: Self-reported prolonged abstinence (primary outcome) will be verified by cotinine assay. Saliva samples will be collected from participants who self-report prolonged abstinence. Prolonged abstinence is defined as continued abstinence from smoking beginning at 2 weeks post-quit.
Time Frame: 6 month follow up
Population: 5 participants were withdrawn from analyses because they were lost to contact before study completion. One was withdrawn by the PI because he couldn't perform study procedures. Two participants didn't self-report abstinence, so bioverification was not completed.
Measure: Count of Participants; unit: Participants
Arm/Group | STEP UP
Number analyzed (Participants) | 3
Participants | 0

3. Primary Outcome: Number of Participants Who Self-report Prolonged Abstinence From Smoking
Description: as for outcome 1
Time Frame: 3 month follow up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | STEP UP
Number analyzed (Participants) | 5
Participants | 0

4. Primary Outcome: Number of Participants Whose Prolonged Abstinence is Bio-verified
Description: as for outcome 2
Time Frame: 3 month follow up
Population: 5 participants were withdrawn from analyses because they were lost to contact before study completion. One was withdrawn by the PI because he couldn't perform study procedures. No participants reported prolonged abstinence, so bioverification wasn't completed.
Arm/Group | STEP UP
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Who Self-report 7 Day Point Prevalence Abstinence From Smoking
Description: 7-day point prevalence abstinence is defined as no smoking in the prior 7 days.
Time Frame: 6 month follow up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | STEP UP
Number analyzed (Participants) | 5
Participants | 0

6. Secondary Outcome: Number of Participants Who Report 30 Day Point Prevalence Abstinence From Smoking
Description: 30-day point prevalence abstinence is defined as no smoking in the prior 30 days.
Time Frame: 6 month follow up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | STEP UP
Number analyzed (Participants) | 5
Participants | 0

7. Secondary Outcome: Number of Participants Who Report 7 Day Point Prevalence Abstinence From Smoking
Description: 7-day point prevalence abstinence is defined as no smoking in the prior 7 days.
Time Frame: 3 month follow up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | STEP UP
Number analyzed (Participants) | 5
Participants | 0

8. Secondary Outcome: Number of Participants Who Report 30 Day Point Prevalence Abstinence From Smoking
Description: 30-day point prevalence abstinence is defined as no smoking in the prior 30 days.
Time Frame: 3 month follow up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | STEP UP
Number analyzed (Participants) | 5
Participants | 0

9. Secondary Outcome: Change in Physical Activity From Baseline to 3-month Follow-up as Measured by the Stanford 7-day Physical Activity Recall (PAR) Scale.
Description: Participants will be interviewed about the amount of time spent in light, moderate, and hard physical activity during the past 7 days. Total number of days of moderate and hard exercise in last 7 days will be compared to self-reported values at baseline (i.e., # of days of exercise in past 7 days at 3-month follow-up minus # of days of exercise in past 7 days at baseline).
Time Frame: baseline and 3 month follow up
Population: Data are only available for two participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | STEP UP
Number analyzed (Participants) | 2
days | -3 (4.24)

10. Secondary Outcome: Change in the Number of Days in Which Smoked Compared to Pre-quit Use
Description: Participants will self-report number of days smoked in the past 30 days and this will be compared to self-reported number of days smoked in 30 days prior to quit.
Time Frame: 3 month follow up
Population: These data were only available for one participant.
Measure: Number; unit: days
Arm/Group | STEP UP
Number analyzed (Participants) | 1
days | 0

11. Secondary Outcome: Change in Number of Cigarettes Smoked Per Week Compared to Pre-quit
Description: Self-reported number of cigarettes smoked each day in past 7 days; this will be compared to self-reported amount smoked in week prior to quit date
Time Frame: 3 month follow up
Population: Only one participant completed the timeline follow-back procedure at 3 months
Measure: Number; unit: cigarettes
Arm/Group | STEP UP
Number analyzed (Participants) | 1
cigarettes | -22

12. Secondary Outcome: Number of Quit Smoking Attempts
Description: Participants will self-report the number of quit attempts they've had since baseline.
Time Frame: 3 month follow up
Population: These data were only available for 2 participants.
Measure: Mean (Standard Deviation); unit: quit attempts
Arm/Group | STEP UP
Number analyzed (Participants) | 2
quit attempts | 4.5 (0.7)

ADVERSE EVENTS:
Time Frame: 6 months
Description: n/a; We utilized clinicaltrials.gov definitions.
Arm/Group | STEP UP
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Several participants had early termination. For appropriate outcomes, intent-to-treat analyses were used, wherein missing=presumed smoking.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT02873754/Prot_SAP_000.pdf